CLINICAL TRIAL: NCT00962299
Title: Effectiveness of Inhaled Corticosteroids in Preschool Children Following Hospital Admission for Acute Dyspnea and Wheeze
Brief Title: Effectiveness of Inhaled Corticosteroids in Preschool Children With Acute Dyspnea and Wheeze
Acronym: ICS@ADP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment was unsuccesfull, only 7 patient have been included untill 2012
Sponsor: Princess Amalia Children's Clinic (Other)
Responsible Party: Principal Investigator, Jolita Bekhof, MD, Pediatrician, Princess Amalia Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL26689.075.09
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Wheezing; Dyspnea
Keywords: Child; Wheezing; Dyspnea; Inhaled corticosteroids
MeSH Terms: conditions — Respiratory Sounds; Dyspnea | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beclomethasone (Active Comparator): Inhaled corticosteroids
  Interventions: Drug: Beclomethasone
- Placebo (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Beclomethasone — Beclometasone 100 ug b.i.d. by metered dose inhaler with spacer for 6 months
  Other Names: Qvar
  Arms: Beclomethasone
Drug: Placebo — Placebo once a day by metered dose inhaler with spacer for 6 months
  Arms: Placebo

SUMMARY:
The aim of the study is to investigate whether inhaled corticosteroids after a first hospital admission for acute dyspnea and wheeze is effective in reducing subsequent episodes of these complaints in children aged 1 to 4 years.

DETAILED DESCRIPTION:
Symptoms of dyspnea and wheeze occur frequently in young children with a cumulative incidence of 33% before the age of 3 and up to 50% by the age of 6 years. Most wheezing episodes in preschool children are associated with viral upper respiratory tract infections (episodic viral wheeze). The majority of children with episodic viral wheeze have become asymptomatic by the age of 6 years. About one in three preschool children with recurrent wheeze continue to wheeze after the age of six years, and these children are usually diagnosed with asthma.

Two clinical phenotypes of recurrent wheezing in preschool children can be distinguished. Children with episodic viral wheeze only wheeze with viral upper respiratory tract infections and are symptom free in between episodes. A minority of children wheeze during upper respiratory tract infection and with other trigger factors (such as smoke, fog, exercise) and this is defined as multiple trigger wheeze.

Inhaled corticosteroids (ICS) have been shown to be effective in preschool children with multiple trigger wheeze, but the effect is smaller than that in older children. This justifies a more critical approach towards such therapy, for example by prescribing a trial of ICS for a period of 3 months and evaluating the effect afterwards. Little research has been performed on the effect of ICS in preschool children with episodic viral wheeze. A high dose of ICS (>1600 ug/d) during an acute episode of dyspnea and wheezing has been shown to be effective, but in a number of small clinical trials maintenance treatment with ICS did not have an effect on the number and severity of episodes of viral wheezing. Contradictory results have been published about the effect of ICS in infants and preschool children with Respiratory Syncytial Virus bronchiolitis. Some studies showed a reduction of wheezing episodes after RSV bronchiolitis in children treated with ICS, two other studies did not show any positive effect.

Prescribing ICS in preschool children can result in adverse effects such as a reduced height growth. Because of the lack of evidence of effect of ICS in episodic viral wheeze, guidelines advise a critical approach towards prescribing ICS in episodic viral wheeze.

ELIGIBILITY:
Inclusion Criteria:

* Children that are admitted to the paediatric ward of the Isala Klinieken in Zwolle for the first time with acute dyspnea and wheezing
* Age 1 - 4 years
* Child and parents must understand the Dutch language well
* Informed consent

Exclusion Criteria:

* Previous use of medication different than short-acting β2-agonists before hospital admission
* Proven RSV bronchiolitis
* Crackles during auscultation of the lungs (suggestive for RSV bronchiolitis)

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Number of unscheduled doctor visits for dyspnea and wheezing | One and a half, 3, 6 and 9 months after discharge.

SECONDARY OUTCOMES:
PACQLQ scores and the use of additional asthma medication | One and a half, 3, 6 and 9 months after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: N Doornebal, MD, Principal Investigator — Princess Amalia Children's Clinic; J Bekhof, MD, Study Director — Princess Amalia Children's Clinic; P LP Brand, MDPhD, Study Director — Princess Amalia Children's Clinic
Locations (1):
- Princess Amalia Children's Clinic, Zwolle, Overijssel, Netherlands

REFERENCES:
- [Result] Martinez FD, Wright AL, Taussig LM, Holberg CJ, Halonen M, Morgan WJ. Asthma and wheezing in the first six years of life. The Group Health Medical Associates. N Engl J Med. 1995 Jan 19;332(3):133-8. doi: 10.1056/NEJM199501193320301. PMID 7800004
- [Result] Hess J, De Jongste JC. Epidemiological aspects of paediatric asthma. Clin Exp Allergy. 2004 May;34(5):680-5. doi: 10.1111/j.1365-2222.2004.1961.x. No abstract available. PMID 15144456
- [Result] Brand PL, Baraldi E, Bisgaard H, Boner AL, Castro-Rodriguez JA, Custovic A, de Blic J, de Jongste JC, Eber E, Everard ML, Frey U, Gappa M, Garcia-Marcos L, Grigg J, Lenney W, Le Souef P, McKenzie S, Merkus PJ, Midulla F, Paton JY, Piacentini G, Pohunek P, Rossi GA, Seddon P, Silverman M, Sly PD, Stick S, Valiulis A, van Aalderen WM, Wildhaber JH, Wennergren G, Wilson N, Zivkovic Z, Bush A. Definition, assessment and treatment of wheezing disorders in preschool children: an evidence-based approach. Eur Respir J. 2008 Oct;32(4):1096-110. doi: 10.1183/09031936.00002108. PMID 18827155
- [Result] Kaditis AG, Winnie G, Syrogiannopoulos GA. Anti-inflammatory pharmacotherapy for wheezing in preschool children. Pediatr Pulmonol. 2007 May;42(5):407-20. doi: 10.1002/ppul.20591. PMID 17358042
- [Result] McKean M, Ducharme F. Inhaled steroids for episodic viral wheeze of childhood. Cochrane Database Syst Rev. 2000;2000(2):CD001107. doi: 10.1002/14651858.CD001107. PMID 10796596
- [Result] King VJ, Viswanathan M, Bordley WC, Jackman AM, Sutton SF, Lohr KN, Carey TS. Pharmacologic treatment of bronchiolitis in infants and children: a systematic review. Arch Pediatr Adolesc Med. 2004 Feb;158(2):127-37. doi: 10.1001/archpedi.158.2.127. PMID 14757604
- [Result] Hesselmar B, Adolfsson S. Inhalation of corticosteroids after hospital care for respiratory syncytial virus infection diminishes development of asthma in infants. Acta Paediatr. 2001 Mar;90(3):260-3. PMID 11332164
- [Result] Kajosaari M, Syvanen P, Forars M, Juntunen-Backman K. Inhaled corticosteroids during and after respiratory syncytial virus-bronchiolitis may decrease subsequent asthma. Pediatr Allergy Immunol. 2000 Aug;11(3):198-202. doi: 10.1034/j.1399-3038.2000.00068.x. PMID 10981531
- [Result] Reijonen T, Korppi M, Kuikka L, Remes K. Anti-inflammatory therapy reduces wheezing after bronchiolitis. Arch Pediatr Adolesc Med. 1996 May;150(5):512-7. doi: 10.1001/archpedi.1996.02170300066013. PMID 8620234
- [Result] Guilbert TW, Morgan WJ, Zeiger RS, Mauger DT, Boehmer SJ, Szefler SJ, Bacharier LB, Lemanske RF Jr, Strunk RC, Allen DB, Bloomberg GR, Heldt G, Krawiec M, Larsen G, Liu AH, Chinchilli VM, Sorkness CA, Taussig LM, Martinez FD. Long-term inhaled corticosteroids in preschool children at high risk for asthma. N Engl J Med. 2006 May 11;354(19):1985-97. doi: 10.1056/NEJMoa051378. PMID 16687711
- [Result] Ducharme FM, Lemire C, Noya FJ, Davis GM, Alos N, Leblond H, Savdie C, Collet JP, Khomenko L, Rivard G, Platt RW. Preemptive use of high-dose fluticasone for virus-induced wheezing in young children. N Engl J Med. 2009 Jan 22;360(4):339-53. doi: 10.1056/NEJMoa0808907. PMID 19164187
- [Result] Raat H, Bueving HJ, de Jongste JC, Grol MH, Juniper EF, van der Wouden JC. Responsiveness, longitudinal- and cross-sectional construct validity of the Pediatric Asthma Quality of Life Questionnaire (PAQLQ) in Dutch children with asthma. Qual Life Res. 2005 Feb;14(1):265-72. PMID 15789960
- [Result] Ermers MJ, Rovers MM, van Woensel JB, Kimpen JL, Bont LJ; RSV Corticosteroid Study Group. The effect of high dose inhaled corticosteroids on wheeze in infants after respiratory syncytial virus infection: randomised double blind placebo controlled trial. BMJ. 2009 Mar 31;338:b897. doi: 10.1136/bmj.b897. PMID 19336497